CLINICAL TRIAL: NCT01203683
Title: Attention Training for Major Depressive Disorder
Brief Title: Testing the Effectiveness of a Computer-based Program for Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-09-0004
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Computer-Based Program (Experimental): Putatively therapeutic computer program.
  Interventions: Behavioral: Active computer-based training
- Placebo computer-based program (Placebo Comparator): Inert computer program.
  Interventions: Behavioral: Inert computer training

INTERVENTIONS:
Behavioral: Active computer-based training — 8 sessions across 4 weeks.
  Arms: Active Computer-Based Program
Behavioral: Inert computer training — 8 sessions across 4 weeks.
  Arms: Placebo computer-based program

SUMMARY:
The purpose of this study is to determine whether completing a computer-based program alters changes how the brain processes emotional information and improves symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder

Exclusion Criteria:

* Substance dependence, psychotic disorder, bipolar disorder, schizophrenia, current psychotherapy, medications other than selective serotonin reuptake inhibitors

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | Week 4, Week 9
  Questionnaire to assess depression symptom severity

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-IV diagnoses | Week 9
  Diagnostic interview to assess for presence of Major depressive disorder (MDD).
Neural processing of emotion stimuli | Week 4
  fMRI paradigm to assess neural changes in how individuals processes emotional stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Beevers, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States